CLINICAL TRIAL: NCT06879860
Title: The Effects of 3D Patch Fixation With One Suture Versus no Fixation on Chronic Pain and Recurrence in Patients With Ⅲ Type Inguinal Hernia: A Multicenter Randomized Controlled Trial
Brief Title: The Impact of 3D Patch One-Suture Fixation vs No Fixation on Chronic Pain and Recurrence in Ⅲ Inguinal Hernia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchong Central Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024156
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one-stitch fixation (Experimental)
  Interventions: Procedure: 3D Mesh Single-Suture Fixation
- non-fixation (Active Comparator)
  Interventions: Procedure: 3D mesh Non-FIxation

INTERVENTIONS:
Procedure: 3D Mesh Single-Suture Fixation — 3D mesh fixation in 1 points
  Arms: one-stitch fixation
Procedure: 3D mesh Non-FIxation — 3D mesh fixation with non-flxation
  Arms: non-fixation

SUMMARY:
This study aims to compare the effects of one-stitch fixation and non-fixation of 3D patches on chronic pain and recurrence in type III inguinal hernia. The primary outcome measures include hernia recurrence, chronic pain, etc.

ELIGIBILITY:
Inclusion Criteria:

1. primary inguinal hernia
2. Type III inguinal hernia (internal annulus >3cm)

Exclusion Criteria:

1. Age below 18 years or older than 80. recurrent hernia, incarcerated hernia,strangulated hernia, and other types of hernias.
2. Patients not suitable for general anesthesia.
3. Patients requiring open surgery.
4. patients requiring emergency surgery Loss to follow-up or communication difficulties, or poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrence | 1 month,3 months,6 months and 12 months after surgery
  Hernia recurrence Follow up by physical examination, ultrasonography and telephone at 1 month,3 months,6 months and 12 months after surgery about the rate of hernia recurrence.
Rate of postoperative pain | 6 month
  The visual analog scale (VAS) was adopted for pain evaluation 2 days, 3 months, and 6 months postoperatively. The scale range from 0 to 10, with 0 meaning no pain and 10 meaning the worst pain.

SECONDARY OUTCOMES:
Rate of postoperative complications | 6 month
  Including infection, seroma, hematoma

CONTACTS AND LOCATIONS:
Locations (1):
- Nanchong Central Hospital, Nanchong, Sichuan, China